CLINICAL TRIAL: NCT05257447
Title: Pharmacokinetic and Bioequivalence Comparison of Baclofen and Chlorzoxazone When Administered Individually or Concurrently
Brief Title: Pharmacokinetic and Bioequivalence Comparison of Baclofen and Chlorzoxazone Administered Individually or Concurrently
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Tufts University (Other)
Responsible Party: Principal Investigator, Vikram Shakkottai, Associate Professor of Neurology, Dedman Family Distinguished Chair in Neurological Disease, Vice Chair for Basic Science Research, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU2021-0797
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Pharmacokinetics
Keywords: baclofen; chlorzoxazone; pharmacokinetics
MeSH Terms: interventions — Baclofen; Tablets; Chlorzoxazone

STUDY DESIGN:
Intervention Model Description: The study will have a randomized, single-dose, 3-way crossover design, with at least one week elapsing between the 3 trials of the study. The sequence of administration is based on a randomization code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baclofen 20mg tablet (Experimental): Single oral dose of baclofen, 20 mg
  Interventions: Drug: Baclofen 20 mg Tablet
- Chlorzoxazone 500mg tablet (Experimental): Single oral dose of chlorzoxazone, 500 mg
  Interventions: Drug: Chlorzoxazone 500 mg Tablet
- Baclofen 20 mg tablet and chlorzoxazone 500 mg tablet (Experimental): Concurrent doses of baclofen, 20 mg, and chlorzoxazone, 500 mg
  Interventions: Drug: Baclofen 20mg tablet and Chlorzoxazone 500 mg tablet

INTERVENTIONS:
Drug: Baclofen 20 mg Tablet — Single oral dose given at approximately 8 AM on day of visit, with 6-8 ounces of tap water.
  Arms: Baclofen 20mg tablet
Drug: Chlorzoxazone 500 mg Tablet — Single oral dose given at approximately 8 AM on day of visit, with 6-8 ounces of tap water.
  Arms: Chlorzoxazone 500mg tablet
Drug: Baclofen 20mg tablet and Chlorzoxazone 500 mg tablet — Concurrent single oral dose given at approximately 8 AM on day of visit, with 6-8 ounces of tap water.
  Arms: Baclofen 20 mg tablet and chlorzoxazone 500 mg tablet

SUMMARY:
Combination treatment with baclofen and chlorzoxazone (CHZ) is under investigation for the treatment of spinocerebellar ataxia types 1 and 2. Achievement of therapeutic benefit with this combination approach requires that effective concentrations of both agents reach the systemic circulation, and ultimately reach the intended pharmacologic target. This in turn requires understanding of the clinical pharmacokinetic properties of both drugs when administered individually, as well as knowledge of the extent to which the agents might interact when given concurrently.

Study Objectives:

1. To evaluate the pharmacokinetic properties of baclofen and CHZ when administered as individual entities at separate times, using customary clinical doses.
2. To compare the pharmacokinetic properties, and assess the bioequivalence, of each drug administered separately compared to administration of the two drugs concurrently.
3. To assess adverse events attributed to the two drugs when administered separately or together.

DETAILED DESCRIPTION:
Baclofen has been available for clinical use in the United States since 1977 and is used for the treatment of spasticity arising from a variety of causes. Oral baclofen can be administered in tablet form or as a solution. Comparison of the kinetics of IV and oral baclofen indicates that absolute bioavailability is in the range of 75%. Clearance of S-baclofen, the pharmacologically active enantiomer, occurs mainly by renal excretion of the intact drug. A small fraction of the administered R-enantiomer is also biotransformed by deamination. In individuals with normal renal function, the elimination half-life is in the range of 3 to 6 hours. Clearance is reduced and half-life is prolonged when renal function is impaired. Baclofen pharmacokinetics are linear (dose-independent), in that half-life and clearance are fixed regardless of the administered dose, or duration of treatment.

Chlorzoxazone (CHZ) has been in clinical use since 1988 and is described as a skeletal muscle relaxant. The principal metabolic pathway of CHZ involves hydroxylation by the hepatic enzyme Cytochrome P450-2E1 (CYP2E1), yielding the major metabolite 6-OH-CHZ. As a substrate for the single enzyme isoform CYP2E1, CHZ has become extensively used in drug development and clinical pharmacology as an in vivo probe or index compound to profile human CYP2E1 metabolic phenotype, based on systemic clearance or area under the plasma concentration curve (AUC) after a single test dose. In healthy individuals, the elimination half-life of CHZ falls in the range of 0.7 to 2.0 hours. With this short half-life, a pharmacokinetic study can be completed using a sampling period of 12 hours after a single dose.

The study will have a randomized, single-dose, 3-way crossover design, with at least one week elapsing between the 3 trials of the study. The sequence of administration is based on a randomization code. Venous blood samples are drawn prior to the dose, and at specified time points during 24 hours after the dose. Concentrations of baclofen and/or chlorzoxazone are determined in each sample, and customary pharmacokinetic analyses are used to evaluate kinetic properties, and bioequivalence between individual versus combined administration of the two drugs.

Candidates for participation will come to the study site for an interview and screening evaluation. Screening procedures will include medical history, medication use (including non-prescription and herbal), physical examination, blood hematology and clinical chemistry, blood immunology screen (HIV and hepatitis), urinalysis, urine drug screen, and serum pregnancy test (for potentially childbearing female participants). Screening data for each subject is reviewed by the Principal Investigator through a global evaluation of all information. The PI then decides whether participation would be safe and reasonable. The PI can choose to decline a candidate's approval as a study subject if the available information indicates that participation would be unsafe or inappropriate.

Subjects arrive at the study unit at 7 AM on each of the three study trial days, following an overnight fast. They are provided with a light breakfast on arrival. Peripheral venous sampling access is established via an indwelling catheter, connected to intravenous fluid (D5W or normal saline) at a "keep open" rate. A heparin lock can also be used - this is flushed with dilute heparin (5 Units per mL) after each sample is drawn. Venous blood samples (7 mL each) are drawn from the indwelling catheter into heparinized (green-top) tubes prior to dosage, and at the following post-dosage times: 1, 2, 3, 4, 6, 8, 10, and 12 hours. Subjects return to the study unit at 8 AM the following morning, at which time a 24-hour PK sample and repeat hematology and chemistry is drawn. The PI or designate will conduct a structured interview to evaluate the occurrence of adverse events

Plasma concentrations of baclofen or chlorzoxazone, as appropriate, will be determined by liquid chromatography-mass spectrometry using contemporary methodology which has been validated, and conforms to customary regulatory standards for sensitivity, specificity, replicability, precision, and accuracy. All samples from a given subject's set of 3 trials will be extracted and analyzed on the same day using the same calibration standards by Tufts University.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Ages 18 to 55 years of age
* Ambulatory
* Non-smoker
* No current or past history of significant medical or psychiatric disease
* Not currently taking prescription medications or on a regular or recurrent basis

Exclusion Criteria:

* Non-ambulatory
* Smokers
* Current or past history of significant medical or psychiatric disease
* Currently taking prescription medications or taking on a regular or recurrent basis
* Available information about potential participant indicates that participation would not be safe or appropriate, per PI discretion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Comparison of the maximum measured plasma concentration (Cmax) of baclofen or chlorzoxazone administered separately with baclofen-chlorzoxazone administered concurrently. | Pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
  Compare the pharmacokinetic properties and assess bioequivalence of baclofen and chlorzoxazone administered separately compared to baclofen-chlorzoxazone administered concurrently, determined by liquid chromatography-mass spectrometry. Maximum measured plasma concentration (Cmax) will be reported.
Compare the area Under the Plasma Concentration Versus Time Curve (AUC) of baclofen and chlorzoxazone administered separately with baclofen-chlorzoxazone administered concurrently. | Pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose
  Evaluate the pharmacokinetic properties of baclofen and chlorzoxazone administered individually, determined by liquid chromatography-mass spectrometry with baclofen-chlorzoxazone administered concurrently. Area under the plasma concentration curve until the last non-zero concentration (AUC-last) will be reported.

OTHER OUTCOMES:
Number of adverse events reported as mild, moderate, or severe | Visit 1 Day 1, Visit 1 Day 2, Visit 2 Day 1, Visit 2 Day 2, Visit 3, Day 1, Visit 3 Day 2
  Number adverse events is assessed by structured interview conducted to evaluate the occurrence of adverse events. The intensity/ seriousness of the AE ranges from 1-3, where higher scores indicate worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Shakkottai, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after de-identification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal should direct inquiries to vikram.shakkottai@utsouthwestern.edu. Data requestors may need to sign a data access agreement.

REFERENCES:
- [Background] Agarwal SK, Kriel RL, Cloyd JC, Coles LD, Scherkenbach LA, Tobin MH, Krach LE. A pilot study assessing pharmacokinetics and tolerability of oral and intravenous baclofen in healthy adult volunteers. J Child Neurol. 2015 Jan;30(1):37-41. doi: 10.1177/0883073814535504. Epub 2014 Jul 14. PMID 25028414
- [Background] Schmitz NS, Krach LE, Coles LD, Mishra U, Agarwal SK, Cloyd JC, Kriel RL. A Randomized Dose Escalation Study of Intravenous Baclofen in Healthy Volunteers: Clinical Tolerance and Pharmacokinetics. PM R. 2017 Aug;9(8):743-750. doi: 10.1016/j.pmrj.2016.11.002. Epub 2016 Nov 17. PMID 27867020
- [Background] Simon N, Franchitto N, Rolland B. Pharmacokinetic Studies of Baclofen Are Not Sufficient to Establish an Optimized Dosage for Management of Alcohol Disorder. Front Psychiatry. 2018 Oct 5;9:485. doi: 10.3389/fpsyt.2018.00485. eCollection 2018. PMID 30349489
- [Background] Lal R, Sukbuntherng J, Tai EH, Upadhyay S, Yao F, Warren MS, Luo W, Bu L, Nguyen S, Zamora J, Peng G, Dias T, Bao Y, Ludwikow M, Phan T, Scheuerman RA, Yan H, Gao M, Wu QQ, Annamalai T, Raillard SP, Koller K, Gallop MA, Cundy KC. Arbaclofen placarbil, a novel R-baclofen prodrug: improved absorption, distribution, metabolism, and elimination properties compared with R-baclofen. J Pharmacol Exp Ther. 2009 Sep;330(3):911-21. doi: 10.1124/jpet.108.149773. Epub 2009 Jun 5. PMID 19502531
- [Background] Vlavonou R, Perreault MM, Barriere O, Shink E, Tremblay PO, Larouche R, Pichette V, Tanguay M. Pharmacokinetic characterization of baclofen in patients with chronic kidney disease: dose adjustment recommendations. J Clin Pharmacol. 2014 May;54(5):584-92. doi: 10.1002/jcph.247. Epub 2014 Jan 10. PMID 24414993
- [Background] Court MH, Von Moltke LL, Shader RI, Greenblatt DJ. Biotransformation of chlorzoxazone by hepatic microsomes from humans and ten other mammalian species. Biopharm Drug Dispos. 1997 Apr;18(3):213-26. doi: 10.1002/(sici)1099-081x(199704)18:33.0.co;2-0. PMID 9113344
- [Background] Valicherla GR, Mishra A, Lenkalapelly S, Jillela B, Francis FM, Rajagopalan L, Srivastava P. Investigation of the inhibition of eight major human cytochrome P450 isozymes by a probe substrate cocktail in vitro with emphasis on CYP2E1. Xenobiotica. 2019 Dec;49(12):1396-1402. doi: 10.1080/00498254.2019.1581301. Epub 2019 Jun 19. PMID 30747554
- [Background] Hohmann N, Blank A, Burhenne J, Suzuki Y, Mikus G, Haefeli WE. Simultaneous phenotyping of CYP2E1 and CYP3A using oral chlorzoxazone and midazolam microdoses. Br J Clin Pharmacol. 2019 Oct;85(10):2310-2320. doi: 10.1111/bcp.14040. Epub 2019 Aug 9. PMID 31222796
- [Background] Streetman DS, Bertino JS Jr, Nafziger AN. Phenotyping of drug-metabolizing enzymes in adults: a review of in-vivo cytochrome P450 phenotyping probes. Pharmacogenetics. 2000 Apr;10(3):187-216. doi: 10.1097/00008571-200004000-00001. PMID 10803676
- [Background] Lucas D, Ferrara R, Gonzalez E, Bodenez P, Albores A, Manno M, Berthou F. Chlorzoxazone, a selective probe for phenotyping CYP2E1 in humans. Pharmacogenetics. 1999 Jun;9(3):377-88. doi: 10.1097/00008571-199906000-00013. PMID 10471070
- [Background] Ernstgard L, Warholm M, Johanson G. Robustness of chlorzoxazone as an in vivo measure of cytochrome P450 2E1 activity. Br J Clin Pharmacol. 2004 Aug;58(2):190-200. doi: 10.1111/j.1365-2125.2004.02132.x. PMID 15255802
- [Background] Mishin VM, Rosman AS, Basu P, Kessova I, Oneta CM, Lieber CS. Chlorzoxazone pharmacokinetics as a marker of hepatic cytochrome P4502E1 in humans. Am J Gastroenterol. 1998 Nov;93(11):2154-61. doi: 10.1111/j.1572-0241.1998.00612.x. PMID 9820389
- [Background] He Q, Chhonker YS, McLaughlin MJ, Murry DJ. Simultaneous Quantitation of S(+)- and R(-)-Baclofen and Its Metabolite in Human Plasma and Cerebrospinal Fluid using LC-APCI-MS/MS: An Application for Clinical Studies. Molecules. 2020 Jan 8;25(2):250. doi: 10.3390/molecules25020250. PMID 31936209
- [Background] He J, Li N, Xu J, Zhu J, Yu Y, Chen X, Lu Y. An LC-MS/MS Validated Method for Quantification of Chlorzoxazone in Human Plasma and Its Application to a Bioequivalence Study. J Chromatogr Sci. 2019 Aug 16;57(8):751-757. doi: 10.1093/chromsci/bmz052. PMID 31363741
- [Background] Noe DA. Parameter Estimation and Reporting in Noncompartmental Analysis of Clinical Pharmacokinetic Data. Clin Pharmacol Drug Dev. 2020 Jul;9 Suppl 1:S5-S35. doi: 10.1002/cpdd.810. PMID 32706165
- [Background] Zhao Y, Harmatz JS, Epstein CR, Nakagawa Y, Kurosaki C, Nakamura T, Kadota T, Giesing D, Court MH, Greenblatt DJ. Favipiravir inhibits acetaminophen sulfate formation but minimally affects systemic pharmacokinetics of acetaminophen. Br J Clin Pharmacol. 2015 Nov;80(5):1076-85. doi: 10.1111/bcp.12644. Epub 2015 Jun 8. PMID 25808818
- [Background] Johnson-Agbakwu C, Brown L, Yuan J, Kissling R, Greenblatt DJ. Effects of Flibanserin on the Pharmacokinetics of a Combined Ethinylestradiol/Levonorgestrel Oral Contraceptive in Healthy Premenopausal Women: A Randomized Crossover Study. Clin Ther. 2018 Jan;40(1):64-73. doi: 10.1016/j.clinthera.2017.08.021. Epub 2017 Dec 2. PMID 29198449
- [Background] Greenblatt DJ, Abourjaily PN. Pharmacokinetics and Pharmacodynamics for Medical Students: A Proposed Course Outline. J Clin Pharmacol. 2016 Oct;56(10):1180-95. doi: 10.1002/jcph.732. Epub 2016 May 9. No abstract available. PMID 26987681